CLINICAL TRIAL: NCT07275398
Title: Psychophysical Well-being, Psychological Distress, and Physical Exercise: An Experimental Study in a Sample of University Students.
Brief Title: Experimental Study on Exercise and Well-being in University Students
Acronym: WE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Jessica Dagani, PhD Candidate, Department of clinical and experimental science, University of Brescia, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNIBS_2024_eserciziowellbeing
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: University Students
Keywords: University Students; Physical Exercise; Well-being
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, Control group - Online Stress Management Program (Active Comparator): Participants in the control group (Group 1) completed a brief, online, asynchronous stress management intervention based on the World Health Organization's Doing What Matters in Times of Stress program. The program consists of five self-guided modules grounded in Acceptance and Commitment Therapy principles, providing practical strategies to manage stress in daily life. One new module was released each week over a five-week period.
  Interventions: Behavioral: Stress Management Program
- Group 2, Experimental Group - Physical Exercise Program plus Stress Management program (Experimental): Participants in the Group 2 completed the same online stress management program as the control group (Group 1), combined with a structured physical exercise program. The physical exercise program consisted of group sessions held twice a week for ten consecutive weeks. The training sessions included whole-body workouts combining aerobic and anaerobic free-body exercises. Students could choose among different types of exercise classes offered by the university sports center, all designed to have comparable intensity levels. All sessions were conducted by certified professional trainers, under the supervision of a qualified sports professional to ensure safety and consistency across activities.
  Interventions: Behavioral: Structured physical exercise program; Behavioral: Stress Management Program

INTERVENTIONS:
Behavioral: Structured physical exercise program — The physical exercise program consisted of group sessions held twice a week for ten consecutive weeks. The training sessions included whole-body workouts combining aerobic and anaerobic free-body exercises. Students could choose among different types of exercise classes offered by the university sports center, all designed to have comparable intensity levels. All sessions were conducted by certified professional trainers, under the supervision of a qualified sports professional to ensure safety and consistency across activities.
  Arms: Group 2, Experimental Group - Physical Exercise Program plus Stress Management program
Behavioral: Stress Management Program — brief, online, asynchronous stress management intervention based on the World Health Organization's Doing What Matters in Times of Stress program (WHO, 2020). The program consists of five self-guided modules grounded in Acceptance and Commitment Therapy principles, providing practical strategies to manage stress in daily life. One new module was released each week over a five-week period, and participants were encouraged to complete the exercises included between modules.

SUMMARY:
The goal of this randomized controlled trial is to to evaluate the effectiveness of a structured physical exercise program in improving university students' well-being. The study involves university students who volunteered to participate in a 10-week intervention designed to enhance their physical and psychological well-being.

The main question it aims to answer is: does participation in the structured physical exercise program lead to greater improvements in psychophysical well-being compared to the control group? Researchers will compare the experimental group (Group 2: structured physical activity program + stress management program) with the active control group (Group 1: stress management program only) to determine whether adding structured physical activity components produces additional benefits. Participants in the experimental Group will engage in a 10 week supervised physical activity program, twice a week, provided by the university sports center, and will attend an online asynchronous stress management program including 5 modules and lasting 5 weeks (one module per week).

Participants in the active control group will only attend the online asynchronous stress management program.

Participants of both groups will complete questionnaires at three time points (baseline, post-intervention, and 3-month follow-up) assessing well-being, psychological distress, quality of life, academic motivation and self-efficacy.

ELIGIBILITY:
Inclusion criteria are: (a) being currently enrolled at a the university of Brescia, and (b) having sufficient proficiency in the Italian language. Exclusion criteria are: (a) any physical condition or illness that would prevent or make exercise unsafe, (b) serious physical injuries (e.g., fractures) within the previous six months, and (c) regular engagement in high-intensity physical activity, defined as belonging to the "high" physical activity level according to the International Physical Activity Questionnaire - Short Form (IPAQ-SF, Mannocci et al., 2010), which classifies individuals into three levels of physical activity (low, moderate, and high).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  The GHQ-12 (Goldberg & Blackwell, 1970) served as the primary outcome measure, assessing overall distress and general well-being. Items are rated on a 4-point Likert scale (0 = "Not at all", 3 = "Much more than usual"), and total scores are summed, with higher scores indicating greater distress.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006): a 7-item self-report questionnaire assessing state anxiety symptoms over the past two weeks. Items are rated on a 4-point scale (0 = "Not at all", 3 = "Nearly every day"), and the total score is summed, with higher scores indicating more severe anxiety.
Patient Health Questionnaire-9 | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001): a 9-item instrument widely used for screening and assessing the severity of depressive symptoms. Items are rated on a 4-point scale (0 = "Not at all", 3 = "Nearly every day"), and the total score is summed, with higher scores reflecting more severe depressive symptoms.
Dropout intention | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  Dropout Intention Scale - adapted version (Biasi et al., 2017; De Vincenzo, 2024; Hardre & Reeve, 2003): this 4-item scale measures students' intentions to withdraw from university, assessing the frequency of dropout-related thoughts and intentions. Items are rated on a 5-point Likert scale (1 = "Never", 5 = "Always"), and the mean score represents overall dropout intention, with higher scores indicating stronger intentions.
Perceived Self-Efficacy Scale | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  Perceived Self-Efficacy Scale (SASP; Pastorelli & Picconi, 2001): This 9-item scale assesses students' perceived ability to focus on and manage academic tasks. Items are rated on a 5-point Likert scale (1 = "Not capable at all", 5 = "Fully capable"), and the final score is the mean of all items, with higher scores indicating greater perceived academic self-efficacy.
Academic Motivation Scale | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  Academic Motivation Scale (AMS; Alivernini & Lucidi, 2008): Based on Self-Determination Theory (Vallerand et al., 1992), the adapted AMS assesses students' academic motivation across five subscales: Amotivation, External Regulation, Introjected Regulation, Identified Regulation, and Intrinsic Regulation. Each subscale has four items rated on an 11-point Likert scale (0 = "Not at all true", 10 = "Completely true"), with higher scores indicating stronger endorsement. In this study, only the Amotivation subscale was analyzed separately, while the other four subscales were combined into two composite indices (De Vincenzo, 2024): AMS Controlled Motivation (External + Introjected Regulation) and AMS Autonomous Motivation (Identified + Intrinsic Regulation), each ranging from 0 to 20. Controlled Motivation reflects engagement due to external or internal pressures, whereas Autonomous Motivation reflects engagement driven by personal interest or value
WHOQOL-BREF | The outcome measure is collected before intervention, after intervention and at 3 months follow-up
  The WHOQOL-BREF is a 26-item instrument developed by the World Health Organization to assess overall quality of life. It includes four domains: Physical Health, Psychological Health, Social Relationships, and Environment. Higher scores indicate better perceived quality of life in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Ghilardi, Professor, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Dipartimento di Scienze Cliniche e Sperimentali, Settore di Psicologia, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
An anonymized dataset excluding personally identifiable information and sensitive sociodemographic details. Specific variables to be included will be determined after data cleaning and privacy review.
Time Frame: After publication of the main study results.
Access Criteria: Researchers with a legitimate scientific interest will be able to access the anonymized dataset and supporting documentation. Access will be granted via a public research data repository (e.g., Zenodo), and users will be required to comply with terms of use and appropriately cite the study. Specific variables included in the shared dataset will be determined following data cleaning and privacy review.